CLINICAL TRIAL: NCT02470156
Title: Coalition for a Healthier Community-Utah Women and Girls - Phase II
Brief Title: Coalition for a Healthier Community-Utah Women and Girls - Phase II (UWAG-II)
Acronym: UWAG-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kathleen Digre, MD, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 55195
Record Dates: First submitted 2015-06-03; First posted 2015-06-12 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Obesity; Physical Activity; Diabetes
Keywords: community based participatory research; healthy eating; physical activity; obesity
MeSH Terms: conditions — Obesity; Motor Activity; Diabetes Mellitus | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Intensity Arm (Intervention) (Experimental): Women in the High Intensity (intervention) arm are counseled by a wellness coach and have a group meeting each month. They are also interviewed four times (at baseline, 4 months, 8 months, and 12 months). Women in the high intensity group must have monthly contact with coaches during at least 9 of 12 months via participation in a group activity and/or monthly coaching to receive a "full dose" of the intervention.
  Interventions: Behavioral: High Intensity Arm (Intervention)
- Low Intensity Arm (Comparison) (Active Comparator): Women in the Low Intensity (comparison) arm are interviewed and coached four times during the study (at baseline, 4 months, 8 months, and 12 months).
  Interventions: Behavioral: Low Intensity Arm (Comparison)

INTERVENTIONS:
Behavioral: High Intensity Arm (Intervention) — The high intensity intervention involves monthly wellness coaching, personalized goal setting, and progress tracking in addition to monthly group activities and social support.
  Arms: High Intensity Arm (Intervention)
Behavioral: Low Intensity Arm (Comparison) — The low intensity intervention involves wellness coaching, personalized goal setting, and progress tracking at baseline, 4 months, 8 months, and 12 months.
  Arms: Low Intensity Arm (Comparison)

SUMMARY:
This 12-month randomized trial is designed to evaluate the impact of low intensity (quarterly) versus high intensity (monthly) wellness coaching programs on women's success achieving individual health goals related to active living and healthy eating and changes in these health behaviors over time.

DETAILED DESCRIPTION:
In Utah, rates of obesity are elevated among non-White and Hispanic women (Utah BRFSS Data, 2008-2012). In order to address these disparities, the Coalition for a Healthier Community for Utah Women and Girls (UWAG) was formed to test the effectiveness of interventions for improving health behaviors delivered through community wellness coaches. UWAG is a strong partnership between academic and public health professionals and Community Faces of Utah (CFU), a coalition representing five underserved communities (African, African American, American Indian, Hispanic and, Pacific Islander).

The investigators hypothesize that a wellness coaching program using an evidence-based lifestyle intervention that has been tailored to meet the gender and cultural needs of women from five diverse, often underserved communities, will be significantly more effective in promoting and sustaining behavioral changes than a less intensive wellness coach program. The primary outcome consists of either an increase in the number of fruits and vegetables consumed in an average week and/or in the number of minutes spent doing moderate or vigorous physical activity in an average week, depending on the participant's target goal, at 12 months after enrolling in the study. The investigators view these as proxy measures for obesity prevention and reduction, and are also collecting data to track changes in weight, BMI and waist-to hip ratio throughout the study.

Wellness coaches are lay community members recruited from each of the CFU communities. They received extensive training and support from the UWAG team. After informed consent and completion of baseline study activities, study participants are randomized into intervention (high intensity) and comparison (low intensity) groups. Participants in both groups receive the evidenced-based program, A New Leaf, tailored to address socio-cultural and gender issues and delivered through community wellness coaches from their own communities. Participants in the high-intensity intervention group participate in monthly group activities in addition to monthly wellness coaching sessions. Participants in the low-intensity comparison group participate in health coaching every 4 months. All participants establish their own goals for fruit and vegetable consumption, physical activity, or both. Investigators collect survey and clinical data at baseline, 4, 8, and 12 months after enrolling and once a year after participants complete the intervention. A return on investment analysis will be conducted. The investigators hypothesize that the more intensive program will lead to better outcomes, and they will assess whether the difference in degree of outcomes warrants its additional costs and resources. Survey data are being collected and include information about demographics, health behaviors, goals and progress towards achieving goals, mental health, self-efficacy, and socio-cultural/gender roles/behaviors related to obesity. Clinical data (blood pressure, body mass index, and waist-to hip ratio) are also collected.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as a female
* Self-identifies as a member of one of the 5 target communities: African American, African, American Indian/Alaskan Native, Hispanic/Latina, Pacific Islander
* Subject is age 18 or older
* Not currently participating in the WISEWOMAN Program or another Wellness Coach Program
* Fluent in English, Spanish, or Kirundi
* Willing to be randomized to high versus low intensity wellness coaching program
* Willing to set a goal related to diet or physical activity
* Willing to be followed for 12 months
* Willing to complete interviews and health data collection at baseline, 4, 8, and 12 months

Exclusion Criteria:

* Subject is less than 18 years of age
* Subject is currently participating in a wellness coach program
* Not fluent in English, Spanish, or Kirundi
* Unwilling to be randomized
* Unwilling to be followed for 12 months
* Unwilling to participate in interviews and data collection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 556 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Wellness Coaching Program Effectiveness on Goal Success | 12 months
  The primary outcome is a composite consisting of either an increase in the number of fruits and vegetables consumed in an average week and/ or in the number of minutes spent doing moderate or vigorous physical activity in an average week, depending on the participant's target goal, at 12 months after enrolling in the study.

SECONDARY OUTCOMES:
Health Behaviors of Partners | 12 Months
  Participants will report on changes in the diet and exercise changes of their partners during the 12 month study.
Health Behaviors of Children | 12 Months
  Participants will report on changes in the diet and exercise changes of their children during the 12 month study.
Change in weight | Baseline and 12 Months
Change in Body Mass Index (BMI) | Baseline and 12 Months
Change in waist circumference | Baseline and 12 Months
Change in waist to hip ratio | Baseline and 12 Months
Economic Assessment of the Intervention | 12 Months
  The cost-effectiveness ratio (CER), which assesses the cost per quality-adjusted life year (QALY), will be generated. Gains in QALYs from increased physical activity will be calculated and quantified for women who went from physically inactive to physically active, and from physically inactive to insufficiently active. QALYs will be calculated using weights which represented societal values of health states, and adjusted demographic factors, BMI, medical conditions, and health status.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Digre, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Buder I, Waitzman N, Zick C. The medical costs of low leisure-time physical activity among working-age adults: Gender and minority status matter. Prev Med. 2020 Dec;141:106273. doi: 10.1016/j.ypmed.2020.106273. Epub 2020 Oct 4. PMID 33022316
- [Derived] Buder I, Zick C, Waitzman N, Simonsen S, Sunada G, Digre K. It Takes a Village Coach: Cost-Effectiveness of an Intervention to Improve Diet and Physical Activity Among Minority Women. J Phys Act Health. 2018 Nov 1;15(11):819-826. doi: 10.1123/jpah.2017-0285. Epub 2018 Oct 11. PMID 30309276